CLINICAL TRIAL: NCT02488551
Title: A Computer-Assisted CBT Tool to Enhance Fidelity in CBOCs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Central Arkansas Veterans Healthcare System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Michael A. Cucciare, PhD, Research Health Scientist, Central Arkansas Veterans Healthcare System
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CRE 12-314
Record Dates: First submitted 2015-06-29; First posted 2015-07-02 (Estimated); Results first posted 2022-09-08 (Actual); Last update posted 2022-09-08 (Actual); Status verified 2022-09

CONDITIONS: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- CALM Tools for Living - computer (Experimental): This intervention includes the delivery of CALM via computer
  Interventions: Device: Computer-delivered CALM
- CALM Tools for Living - manual (Active Comparator): This intervention includes the delivery of CALM delivered manual
  Interventions: Other: Manual-delivered CALM

INTERVENTIONS:
Device: Computer-delivered CALM — This intervention includes the delivery of CALM via computer
  Arms: CALM Tools for Living - computer
Other: Manual-delivered CALM — This active comparison condition includes the delivery of CALM via manual
  Arms: CALM Tools for Living - manual

SUMMARY:
Background and Significance: Mental health (MH) providers in VA Community-Based-Outpatient-Clinics (CBOCs) are often located in rural areas and isolated from educational opportunities. Almost half of Veterans now use CBOCs. Studies have shown that the quality of delivery of EBPs (fidelity) impacts clinical outcomes. This study will test a computer-assisted tool (CALM Tools for Living) that increases fidelity to CBT in treating depression and four common anxiety disorders, including PTSD. Although results of a large RCT, the CALM study, suggested that the tool contributed to fidelity to the CBT protocol, this hypothesis has not been tested. This study will test the tool in primarily rural CBOCs in VA VISN16.

Objective: To modify a computer-assisted CBT tool to meet the needs of CBOC MH providers and Veterans, to evaluate the impact on providers' fidelity to the CBT model and clinical outcomes, and to assess how best to support future implementation.

Specific Aims/Hypothesis: (1) Engage CBOC MH providers in modifying the computer-assisted CBT tool such that its content is relevant and acceptable to Veterans and providers. The investigators hypothesize that the modified tool will be acceptable to both Veterans and providers. (2) Compare MH provider fidelity to CBT and clinical outcomes among providers who used the tool and those who did not. The investigators hypothesize that clinicians who use the tool will have a higher fidelity to CBT and clinical outcomes among patients will be superior. (3) Prepare for future implementation of the tool in the VA.

Methodology: This study will use a Type III hybrid effectiveness design. Methods common to the field of Instructional Design and Technology (IDT) will be used to modify the tool. Thirty-four CBOC MH providers will be trained in CBT and randomized to use the tool or not. Both groups will receive external facilitation to encourage the full implementation of CBT into practice on the clinic level. MH providers will treat 10 patients each. Patients will be assessed at baseline, 3, 6, and 12 months. Provider fidelity to the CBT protocol will be measured, and finally, a tool kit for future implementation of the tool will be disseminated.

Impact: The investigators expect the intervention to improve the technical quality of MH treatment in CBOCs and improve clinical outcomes among Veterans.

DETAILED DESCRIPTION:
Power analysis for primary outcome We aimed to recruit a total sample of 34 (17 per condition) providers to achieve a statistical power of 0.94 for analysis comparing our primary outcome of CBT fidelity between the two conditions. We used a general linear mixed model to account for patients clustered within the same providers and a type I error rate of .05. This initial sample size was also determined by assuming an effect size of 1.0 (1.3 point difference on a scale of CBT fidelity; 5.3 of 6 for the computer condition versus 4 of 6 for manual condition), a medium intraclass correlation of 0.5, and four patients per provider.

A total of 16 of 32 clinicians self-selected to provide audiotaped sessions that were assessed for fidelity. Assuming an effect size of 1.0 for condition on the fidelity outcome, an intraclass correlation of 0.5, four participants per provider, and a type I error rate of .05, our statistical power for comparing our primary outcome of fidelity between conditions using general linear mixed model is 0.65.

Statistical analysis For the primary outcome of providers' CBT fidelity, descriptive statistics were calculated for the entire sample and by session. The association between condition and the outcome of fidelity was examined using a general linear mixed model to account for Veteran participants clustered within providers. The treatment session and strata variables were also included in the model.

For the patient-level secondary outcomes, bivariate analysis was performed using generalized estimating equations due to the clustered structure of Veterans within the same providers. Associations between condition and potential covariates and between outcomes and potential covariates were examined. Covariates with p-values less than 0.10 were included in the multivariate models for associations between condition and outcomes over time. Generalized linear mixed models were used to account for the correlations for patients within providers as well as the correlations of multiple assessments within patients. Gamma distribution was specified for BSI-18 GSI scores after a small rescale for zero value due to its violation of normality and normal distribution was specified for the remaining outcomes as they were approximately normally distributed. All the models included the condition indicator variable, time (for the three interviews), strata, and covariates identified in the bivariate analysis. The covariates associated with condition (gender and primary diagnosis) were included in all the models with the exception of primary diagnosis not being included in the subgroup specific diagnosis group analysis. The covariates associated with the outcomes were also included in the corresponding outcome models. The interaction between condition and time was included in all of the models as hypothesized. General linear mixed models were also fit for disorder specific outcomes for subgroups of Veterans with the corresponding specific disorders as they were approximately normally distributed.

The LS mean differences (or ratios depending on the outcomes) between the two conditions and their corresponding 95% confidence intervals were calculated for evaluating the effect of condition. Similar differences (or ratios) between each follow-up and baseline by each condition and their corresponding 97.5% confidence intervals were also calculated for evaluating the effect of time. A narrower confidence interval (equivalent to a p-value of 0.025) was used to adjust for multiple comparisons. All the analyses were performed using SAS 9.4.

ELIGIBILITY:
Inclusion Criteria:

* Patients will be considered eligible if they:

  1. plan to continue to receive mental health care at the CBOC
  2. have depression, PTSD, or other anxiety disorder (PD, GAD, SAD)
  3. want to receive CBT specifically
  4. are willing to have their therapy sessions audio-taped
  5. are willing and able to participate in clinical assessments (baseline, 3, 6, and 12 months) by phone.

Exclusion Criteria:

* Patients will be considered ineligible if they

  1. have significant cognitive impairment, are in crisis (e.g., suicidal)
  2. are dependent on alcohol or drugs (substance abuse is allowed)
  3. have previously completed a course of CBT or CPT treatment (patients who have previously had only one or two sessions of CBT or CPT will be allowed), or (4) have a comorbid diagnosis of schizophrenia or bipolar disorder.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 167 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

REFERENCES:
- [Derived] Cucciare MA, Curran GM, Craske MG, Abraham T, McCarthur MB, Marchant-Miros K, Lindsay JA, Kauth MR, Landes SJ, Sullivan G. Assessing fidelity of cognitive behavioral therapy in rural VA clinics: design of a randomized implementation effectiveness (hybrid type III) trial. Implement Sci. 2016 May 10;11:65. doi: 10.1186/s13012-016-0432-4. PMID 27164866

RESULTS

PARTICIPANT FLOW:
Groups:
- CALM Tools for Living - Computer: Computer-delivered CALM: This intervention includes the delivery of CALM by computer
- CALM Tools for Living - Manual: Manual-delivered CALM: This active comparison condition includes the delivery of CALM by manual
- Mental Health Providers; CALM Tools for Living-Computer: Mental health providers randomized to deliver CALM by computer
- Mental Health Providers: CALM Tools for Living-Manual: Mental health providers randomized to delivery CALM by manual
Period: Overall Study
Arm/Group | CALM Tools for Living - Computer | CALM Tools for Living - Manual | Mental Health Providers; CALM Tools for Living-Computer | Mental Health Providers: CALM Tools for Living-Manual
Started | 86 | 49 | 17 | 15
Completed | 81 | 41 | 17 | 15
Not Completed | 5 | 8 | 0 | 0
Not completed — Lost to Follow-up | 4 | 7 | 0 | 0
Not completed — Military Deployment | 1 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Data on age, sex/gender and race/ethnicity were not collected for mental health providers in either condition (computer or manual)
Groups:
- CALM Tools for Living - Computer: Computer-delivered CALM: This intervention includes the delivery of the CALM intervention by computer
- CALM Tools for Living - Manual: Manual-delivered CALM: This active comparison condition includes the delivery of the CALM intervention by manual
- Mental Health Providers: CALM Tools for Living-computer: Mental health providers randomized to deliver CALM by manual (baseline characteristics on these participants were not collected and thus are not reported)
- Mental Health Providers: CALM Tools for Living-Manual: Mental health providers randomized to deliver CALM by computer (baseline characteristics on these participants were not collected and thus are not reported)
- Total: Total of all reporting groups
Arm/Group | CALM Tools for Living - Computer | CALM Tools for Living - Manual | Mental Health Providers: CALM Tools for Living-computer | Mental Health Providers: CALM Tools for Living-Manual | Total
Number analyzed (Participants) | 86 | 49 | 17 | 15 | 167
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Data were not collected for the "Mental Health Providers: CALM Tools for Living-computer" and "Mental Health Providers: CALM Tools for Living-Manual" Arms/Groups.
  years
    number analyzed (Participants) | 86 | 49 | 0 | 0 | 135
    (all) | 43.20 (12.35) | 44.63 (14.56) |  |  | 43.72 (13.16)
Sex/Gender, Customized [Number; unit: participants] — Population: Data were not collected for the "Mental Health Providers: CALM Tools for Living-computer" and "Mental Health Providers: CALM Tools for Living-Manual" Arms/Groups.
  participants
    Sex : Male: number analyzed (Participants) | 86 | 49 | 0 | 0 | 135
    Sex : Male | 60 | 39 |  |  | 99
    Sex : Female: number analyzed (Participants) | 86 | 49 | 0 | 0 | 135
    Sex : Female | 26 | 10 |  |  | 36
Race/Ethnicity, Customized [Number; unit: participants] — Population: Data were not collected for the "Mental Health Providers: CALM Tools for Living-computer" and "Mental Health Providers: CALM Tools for Living-Manual" Arms/Groups.
  participants
    Hispanic: number analyzed (Participants) | 86 | 49 | 0 | 0 | 135
    Hispanic | 15 | 21 |  |  | 36
    Other: number analyzed (Participants) | 86 | 49 | 0 | 0 | 135
    Other | 6 | 6 |  |  | 12
    Black: number analyzed (Participants) | 86 | 49 | 0 | 0 | 135
    Black | 14 | 5 |  |  | 19
    White: number analyzed (Participants) | 86 | 49 | 0 | 0 | 135
    White | 51 | 17 |  |  | 68
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 86 | 49 | 17 | 15 | 167

OUTCOME MEASURES:

1. Primary Outcome: CBT Treatment Fidelity (a Rating Indicating Provider Overall Competence in Delivering the Intervention)
Description: Fidelity was defined as providers' overall competence in delivering the VA CALM protocol, for each rated session (i.e., How skilled was the mental health provider in delivering the information in this section?), rated on a Likert scale of 0 to 6 (higher scores indicate greater fidelity).
Time Frame: 6 months
Population: Participants for this outcome were 32 mental health providers (17 randomized to the computer condition and 15 randomized to the manual condition).We used stratified sampling to randomly select 19% (68/368; 32 and 36 audiotaped treatment sessions in the manual and computer conditions, respectively) of the audiotaped VA CALM sessions across sessions. We pre-specified to report only partial data for this outcome due to resource constraints.
Measure: Mean (Standard Deviation); unit: scores on a scale
Units Other Than Participants: therapy (audio) tapes
Arm/Group | CALM Tools for Living - Computer | CALM Tools for Living - Manual
Number analyzed (Participants) | 17 | 15
Number analyzed (therapy (audio) tapes) | 36 | 32
scores on a scale | 3.99 (.86) | 3.23 (.88)

2. Secondary Outcome: General Mental Health Symptoms (Brief Symptoms Inventory)
Description: The BSI-18 is designed to measure general psychological distress and consists of three six-item subscales (somatization, anxiety, and depression). Respondents are asked to indicate, using a 5-point Likert scale, how much they have been bothered by each symptom over the past week. All 18-items can be summed to derive a total score or GSI score which is an indicator of overall level of psychological distress. GSI scores can range from 0-72, with higher scores representing worse outcomes.
Time Frame: 6-months
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | CALM Tools for Living - Computer | CALM Tools for Living - Manual
Number analyzed (Participants) | 81 | 41
scores on a scale | 19.30 (12.62) | 22.10 (15.53)

3. Secondary Outcome: General Mental Health Symptoms (Short-Form-12 Mental Health Composite)
Description: The SF-12 was designed to measure physical and mental health of persons in the United States, with all items weighted and summed to construct summary scores representing both aspects of overall health.
  Only the mental health composite was used in the present study. Total scores are converted to z-scores and can range from 0-50 with higher scores indicating better mental health functioning.
Time Frame: 6-months
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | CALM Tools for Living - Computer | CALM Tools for Living - Manual
Number analyzed (Participants) | 81 | 41
scores on a scale | 35.53 (6.28) | 35.73 (6.94)

4. Secondary Outcome: Generalized Anxiety Disorder Symptoms
Description: The Generalized Anxiety Disorder-7(GAD-7) is a reliable and valid assessment of GAD symptoms. Participants indicate how bothered (0=not at all, 3=nearly every day) they have been by anxiety symptoms (e.g., trouble relaxing) over the past two weeks. A sum of the GAD-7 scores was used as the outcome. Scores can range from 0-21 with higher scores indicating more anxiety.
Time Frame: 6-months
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | CALM Tools for Living - Computer | CALM Tools for Living - Manual
Number analyzed (Participants) | 81 | 41
scores on a scale | 9.88 (5.81) | 12.00 (5.51)

5. Secondary Outcome: PTSD Symptoms
Description: The Posttraumatic Stress Disorder Checklist for the Diagnostic and Statistical Manual for Mental Disorders (Fifth Edition) was used to assess symptoms of PTSD. Participants are asked to indicate how much they have been bothered (0=not at all, 4=extremely) by each item (e.g., feeling distant or cutoff from other people). A sum of the items on this measure was used for the outcome. Scores can range from 0-80 with higher scores indicating more PTSD symptoms.
Time Frame: 6-months
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | CALM Tools for Living - Computer | CALM Tools for Living - Manual
Number analyzed (Participants) | 81 | 41
scores on a scale | 42.57 (17.09) | 46.00 (17.34)

6. Secondary Outcome: Depression Symptoms
Description: The Patient Health Questionnaire (PHQ-9) was used to measure the severity of depression symptoms. The PHQ-9 is a valid measure for assessing how often participants have been bothered (0=not at all, 3=nearly every day), in the past two weeks, by depression symptoms (e.g., feeling tired or having little energy). A sum of the items on this measure was used for the outcome. Scores can range from 0-27 with higher scores indicating more depression symptoms.
Time Frame: 6-months
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | CALM Tools for Living - Computer | CALM Tools for Living - Manual
Number analyzed (Participants) | 81 | 41
scores on a scale | 13.32 (6.99) | 12.33 (5.85)

ADVERSE EVENTS:
Time Frame: 6-months
Description: All participants were monitored for any adverse risks (serious, and not serious) associated with study participation.
Groups:
- Mental Health Providers; CALM Tools for Living-Computer: This arm includes mental health providers assigned to deliver CALM by computer
- Mental Health Providers; CALM Tools for Living-Manual: This arm includes mental health providers assigned to deliver CALM by manual
Arm/Group | CALM Tools for Living - Computer | CALM Tools for Living - Manual | Mental Health Providers; CALM Tools for Living-Computer | Mental Health Providers; CALM Tools for Living-Manual
All-Cause Mortality (participants affected / at risk) | 0/81 | 0/41 | 0/17 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/81 | 0/41 | 0/17 | 0/15
Other Adverse Events (participants affected / at risk) | 0/81 | 0/41 | 0/17 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-01): https://cdn.clinicaltrials.gov/large-docs/51/NCT02488551/Prot_SAP_000.pdf